CLINICAL TRIAL: NCT06647836
Title: Exploration of the Treatment Trajectory and Drug Resistance Mechanism of Immunotherapy Combined With Chemotherapy in Patients With Advanced Lung Squamous Carcinoma
Brief Title: The Therapeutic Effect of Immunotherapy in Patients With Advanced Lung Squamous Carcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Yang Jin, deputy dean, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: XHJY20240908
Record Dates: First submitted 2024-09-11; First posted 2024-10-18 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Squamous Cell Lung Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples and tumor tissues will be retained.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- untreated sq-NSCLC patients: Patients diagnosed with sq-NSCLC for the first time
  Interventions: Other: Efficacy observation
- sq-NSCLC patients treated with immunotherapy for -2-3 cycles: sq-NSCLC patients treated with immunotherapy combined with or without chemotherapy as first-line treatment for 2-3 cycles.
  Interventions: Other: Efficacy observation
- sq-NSCLC patients receiving immunotherapy with poor efficacy: sq-NSCLC patients treated with immunotherapy combined with or without chemotherapy as first-line treatment and experience disease progression within six months.
  Interventions: Other: Efficacy observation
- sq-NSCLC patients receiving immunotherapy with good efficacy: sq-NSCLC patients treated with immunotherapy combined with or without chemotherapy as first-line treatment and having progression-free survival longer than six months.
  Interventions: Other: Efficacy observation

INTERVENTIONS:
Other: Efficacy observation — Observation about the efficacy of sq-NSCLC patients receiving immunotherapy combined with or without chemotherapy as first-line treatment.

SUMMARY:
The aim of this observational study is to investigate the treatment trajectory of immunotherapy in patients with squamous non-small cell lung cancer (sq-NSCLC). The primary objective is to identify potential indicators that can predict the efficacy of immunotherapy and explore strategies to prolong its effectiveness in sq-NSCLC patients. Biological specimens and medical imaging data will be collected from patients already receiving immunotherapy as a first-line treatment, and follow-up will be conducted to analyze prognosis based on different patterns.

DETAILED DESCRIPTION:
The medical imaging data will be collected retrospectively and prospectively and the blood samples and tumor tissues will be collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sq-NSCLC;
* Receiving immunotherapy combined with or without chemotherapy as first-line treatment;
* ≥ 18 years and ≤ 80 years old;
* No previous treatment in the lungs or any other organ.

Exclusion Criteria:

* History of cancer treatment;
* History of other malignant tumors;
* Irregular treatment or poor compliance;
* Incomplete clinical information or lost to follow-up.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2021 to December 2025, about 1000 patients with sq-NSCLC receiving immunotherapy combined with or without chemotherapy as first-line treatment will be enrolled in this cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | A two-year period after starting treatment (Regular follow-up every three months after receiving immunotherapy combined with or without chemotherapy as first-line treatment)
  The time of disease progression is evaluated according to the Response Evaluation Criteria in Solid Tumors, version 1.1.

SECONDARY OUTCOMES:
Overall survival | A three-year period after starting treatment (Regular follow-up every six months after receiving immunotherapy combined with or without chemotherapy as first-line treatment)
  The survival time aftering receiving immunotherapy combined with or without chemotherapy as first-line treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xueyun Tan, MD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Yang Jin, PHD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical college, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No